CLINICAL TRIAL: NCT05785299
Title: Evaluation of the Outcome of Clinical or Home Introduction of Milk in Children with Non-IgE-mediated Cow's Milk Allergy (ENIGMA Trial)
Brief Title: Clinical Versus Home Introduction of Milk in Children with Non-IgE-mediated Cow's Milk Allergy
Acronym: ENIGMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ABR 83741
Record Dates: First submitted 2023-02-24; First posted 2023-03-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cow Milk Allergy; Food Allergy
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double blind placebo controlled challenge test (Active Comparator): Introduction of cow's milk by means of an adjusted double blind placebo controlled challenge test
  Interventions: Diagnostic Test: Cow's milk; Diagnostic Test: Placebo
- Home introduction test (Active Comparator): Introduction of cow's milk by means of a standardized schedule
  Interventions: Diagnostic Test: Home introduction

INTERVENTIONS:
Diagnostic Test: Cow's milk — clinical introduction of cow's milk
  Other Names: Oral food challenge test
  Arms: Double blind placebo controlled challenge test
Diagnostic Test: Placebo — clinical introduction of placebo
  Other Names: Oral food challenge test
  Arms: Double blind placebo controlled challenge test
Diagnostic Test: Home introduction — home introduction of cow's milk
  Arms: Home introduction test

SUMMARY:
There are a lot of parents who believe that their child may not tolerate cow's milk because they develop symptoms such as redness of the skin or they may vomit. It is not always easy to find out if these infants should indeed avoid drinking cow's milk or that the symptoms are caused by something else, for instance because they have a viral illness. The goal of the investigators is to find out if cow's milk should be introduced in the hospital or if it can also be advised to perform the introduction at home to determine if an infant can drink cow's milk without developing symptoms. Half of the participants will drink cow's milk in the hospital. This test is performed on two days. On one of the days cow's milk will be offered. On the other day a look-alike substance is offered. The other half of the participants will drink cow's milk at home by starting to drink a little bit of milk and in a few steps drink a normal bottle of cow's milk. The main question is whether both tests can be used to find out if an infant can drink cow's milk without developing symptoms.

DETAILED DESCRIPTION:
Cow's milk allergy (CMA) is the most common food allergy among infants. CMA can be divided into immunoglobin E (IgE) and non-IgE-mediated allergy. In case of IgE-mediated allergy, symptoms occur within two hours after ingestion, and are potentially life-threatening. In patients without sensitisation, symptoms may occur up to 48 hours after ingestion and predominantly affect the gastrointestinal tract and skin. The gold standard to diagnose a cow's milk allergy is to perform a double-blind placebo controlled food challenge (DBPCFC). Determination of DBPCFC outcome for non-IgE-mediated allergy can be challenging due to delayed presentation of symptoms after the DBPCFC has been performed. Furthermore, in the majority of infants with non-IgE-mediated cow's milk allergy, symptoms are mild and therefore introduction under medical supervision is superfluous. To date, there is no validated diagnostic to confirm a diagnosis of non-IgE-mediated cow's milk allergy and potential over diagnosis is due to the overlap of symptoms with other common diseases in infants.

The aim of this study is to compare the outcome of an adjusted DBPCFC and introduction at home of cow's milk for children with a suspected non-IgE-mediated cow's milk allergy

Patients with a suspected cow's milk allergy will be randomized to a DBPCFC or home introduction of cow's milk after sensitisation for cow's milk has been excluded and parents have not reported severe symptoms during introduction of cow's milk. Outcome of both introduction methods will be based on predefined criteria. For patients with a negative outcome of the test unrestricted exposure to cow's milk is recommended. In case of a positive outcome, parents are recommended to gradually increase the amount of cow's milk in their child's diet by means of the "milk ladder". During regular follow-up visits the investigators will inquire whether introduction of cow's milk is successful and if needed motivate parents to continue further introduction. Number of all consultations will be registered.

ELIGIBILITY:
Inclusion Criteria:

* maximum age of eighteen months;
* suspected to be allergic for cow's milk (based on medical history);

Exclusion Criteria:

* children older than the age of eighteen months;
* sensitised for cow's milk (i.e. SPT >3mm (in combination with positive control ≥3mm) or specific IgE >0.35 kU/L)
* patient suffers from acute (i.e. within one hour after cow's milk had been eaten) and moderate-severe IgE-mediated symptoms after ingestion of cow's milk
* patient suffers from symptoms according to the FPIES criteria after ingestion of cow's milk
* patient uses beta blockers and/or prednisolone;
* patient suffers from uncontrolled respiratory symptoms or severe eczema or a chronic condition because of which the patients cannot be included as judged by the treating physician;
* parents are unable to adequately report the occurrence of possible symptoms (e.g. insufficient language proficiency).

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a positive or negative test | Determined 1 week after start of the test
  Positive (intolerant) or negative (tolerant) outcome of the introduction test

SECONDARY OUTCOMES:
Regular milk consumption | Determined 6 weeks after completion of the test
  Milk consumption is based on normal daily intake for age
Percentage and type of reported symptoms | Determined 6 weeks after completion of the test
  Reported symptoms are classified according to predefined criteria
Healthcare utilisation during the study period | Determined 6 weeks after completion of the test
  Healthcare utilisation is determined by evaluation of the number of physical and telephone consultations

CONTACTS AND LOCATIONS:
Overall Officials: Kamps, MD, PhD, Principal Investigator — Martini Ziekenhuis Groningen
Locations (1):
- Martini Hospital, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and data will be shared upon request
Supporting Information: Study Protocol, CSR
Time Frame: Data will be analysed after all patients have ended the study period.
Access Criteria: Request by mailing principal investigator